CLINICAL TRIAL: NCT05819255
Title: Comprehensive Assessment of Cancer Immunotherapy Response; Investigating the Intent to Change Treatment Decisions Based Upon TRAQinform Immuno Technology
Brief Title: TRAQinform Assessment of Immunotherapy Response
Acronym: AIQ TRAQinform
Status: Completed | Type: Observational
Sponsor: AIQ Solutions (Industry)
Collaborators: National Cancer Institute (NCI) (NIH); Massachusetts General Hospital (Other); University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: AIQ 22-583; 2R44CA257253 (NIH)
Record Dates: First submitted 2023-04-06; First posted 2023-04-19 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Other: Non-Interventional — This prospective, non-interventional clinical study will enroll patients with metastatic melanoma, who have been selected by their oncologist to receive standard of care dual-agent immunotherapy and monitored for treatment response using SOC FDG PET/CTs.
  The primary objective of this clinical study is to investigate intent to change treatment decisions after the addition of treatment response information from the TRAQinform Immuno technology.

SUMMARY:
The intent of this study is to evaluate the actionable information output from the TRAQinform Immuno technology in a prospective, non-interventional clinical study. Subjects with metastatic melanoma treated with standard of care (SOC) dual-agent immunotherapy will be enrolled. Subjects will receive SOC immunotherapy monitored for treatment response with FDG PET/CT's at baseline (SOC), after 3-4 weeks of treatment (non-SOC) and 12 at weeks of treatment (SOC).

DETAILED DESCRIPTION:
This prospective, non-interventional clinical study will enroll patients with metastatic melanoma, who have been selected by their oncologist to receive standard of care (SOC) dual-agent immunotherapy and monitored for treatment response using SOC FDG PET/CTs.

The primary objective of this clinical study is to investigate intent to change treatment decisions after the addition of treatment response information from the TRAQinform Immuno technology. For each subject, FDG PET/CT #1, #2 and #3 will be transmitted to AIQ Solutions (Madison, WI) for treatment response analysis using TRAQinform Immuno, a software technology that identifies, matches and quantifies metastatic cancer regions of interest. A TRAQinform Immuno report will be returned to the oncology/nuclear medicine paired investigator teams, after the first clinical decision point following FDG PET/CT #1 and #2 and again after the second clinical decision point following FDG PET/CT #3. The investigator team at each site will complete an "intent to change" questionnaire for each subject at Data Collection Point #1 and at Data Collection Point #2. The clinical study will evaluate the Data Collection Point questionnaires to help understand the clinical impact of the addition of TRAQinform Immuno analysis into the clinical workflow.

To address the status quo bias of the investigator teams, the TRAQinform Immuno reports for subjects enrolled at each site, including the additional limited data that is necessary to make a treatment decision, will be shared between teams. The first investigator team, without knowledge of the treatment decision made by the second investigator team, will independently answer the Data Collection Point #3 questionnaire and vice versa.

An exploratory objective of this clinical trial is to investigate if treatment effectiveness and adverse events could be detected on FDG PET/CT images at 3-4 weeks of the combination immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of metastatic melanoma and is planned to start or has received one cycle of treatment with standard of care, dual-agent immunotherapy.
* Previous adjuvant anti-PD-I monotherapy is allowed. Patients must be greater than 6 months from the last treatment.
* Previous adjuvant BRAF/MEK therapy is allowed.
* Ability to tolerate 3 FDG PET/CT procedures. One at baseline, prior to the start of the combination immuno therapy, after 3 - 4 weeks of the combination immunotherapy treatment, and at 12 weeks of the combination treatment.
* Estimated life expectancy of greater than 12 months at screening.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2 at screening.
* Deemed suitable for starting standard of care combination immunotherapy for metastatic melanoma.
* Willing and able to provide informed consent for FDG PET/CT imaging.

Exclusion Criteria:

* Any concurrent disease, infection, or comorbid condition that interferes with the ability of the patient to participate in the trial; places the patient at undue risk; or complicates the interpretation of the data, in the opinion of the investigator.
* A second malignancy
* Pregnancy or women who are breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic melanoma.
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2023-06-23 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
To Investigate Intent to Change Treatment Decisions. | 12 weeks
  Treatment response will be analyzed using TRAQinform Immuno Technology which is a software technology that identifies, matches, and quantifies metastatic cancer regions of interest. The clinical study will evaluate investigator questionaries to help understand the clinical impact of the addition of the TRAQinform Immuno analysis into the clinical work flow.

SECONDARY OUTCOMES:
Adverse Events and Treatment Efficacy Prediction | 4 weeks
  To investigate if treatment effectiveness and adverse events can be detected on week 3-4 FDG PET/CT. An additional FDG PET/CT will be obtained on all subjects between weeks three and four to evaluate if TRAQinform Immuno can predict adverse events and treatment effectiveness.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin